CLINICAL TRIAL: NCT02907671
Title: Effectiveness of Ultrasound Guided Corticoanesthetic Injection in Carpal Tunnel Syndrome Comparing Two Different Injection Sites
Brief Title: Effectiveness of Ultrasound Guided Corticoanesthetic Injection in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehabilitace MUDr. Hasan Mezian s.r.o. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2016-09-10; First posted 2016-09-20 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel injection; corticosteroid; ultrasound-guided; musculoskeletal ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): carpal tunnel corticoanesthetic injection between the flexor tendons
  Interventions: Procedure: carpal tunnel corticoanesthetic injection
- Group B (Active Comparator): carpal tunnel corticoanesthetic injection next to the median nerve with hydrodissection
  Interventions: Procedure: carpal tunnel corticoanesthetic injection

INTERVENTIONS:
Procedure: carpal tunnel corticoanesthetic injection — Different Injection Sites (between the flexot tendons or around the median nerve with hydrodissection)
  Other Names: injetion with corticosteroid and local aneshtetics

SUMMARY:
Effectiveness of ultrasound guided corticoanesthetic injection in carpal tunnel syndrome treatment comparing two different injection sites. Single-blind randomized trial.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common nerve entrapment neuropathy. Six placebo-controlled trials with 393 participants proved corticosteroid injection to be effective in symptom relief. However, all injections were palpation-guided. Therefore, the exact injection site was uncertain. Although three studies comparing palpation and ultrasound (US) guided CTS injection showed US superiority, the optimal injection site for the injectate delivery remains unclear. Some authors believe in thinning of the flexor tenosynovium as the mechanism of the median nerve decompression, and therefore recommend injection between the tendons, away from the nerve. Other authors stress the importance of hydrodissection and direct contact of the injectate with the nerve and suggest injection targeting the median nerve. According to our best knowledge, no study comparing different injection sites for a corticosteroid delivery in CTS has been published in English written literature. The objective of this study was to determine the optimal target site for the corticosteroid delivery in CTS injection.

ELIGIBILITY:
Inclusion Criteria:

* primary idiopathic CTS
* symptoms of classic or probable CTS (numbness or tingling in at least 2 of the 4 radial fingers)
* unsuccessful 1-month treatment with wrist splinting
* nerve conduction test results that showed median neuropathy at the wrist

Exclusion Criteria:

* previous steroid injection
* diabetes mellitus,
* thyroid disorder
* inflammatory disease
* polyneuropathy
* current pregnancy
* previous carpal tunnel surgery
* severe illness
* inability to respond to questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | up to 1 year
  pain severity scale

SECONDARY OUTCOMES:
Michigan Hand Outcomes Measure | up to 1 year
  Hand function status
Boston carpal tunnel questionnaire | up to 1 year
  Hand function status
Procedural CAS | up to 1 year
  discomfort during the internetion

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Mezian, M.D., Principal Investigator — Czech Technical University in Prague, Faculty of Biomedical Engineering, Department of Health Care Disciplines and Population Protection, Sportovců 2311, 272 01 Kladno city, Czech Republic
Locations (2):
- Czechia (2):
  - Kamal Mezian, Litoměřice, Czech Republic
  - Kamal Mezian, Litoměřice

IPD SHARING:
Plan to Share IPD: Yes
Publication in the relevant journal

REFERENCES:
- [Result] Mezian K, Bruthans J. Why do local corticosteroid injections work in carpal tunnel syndrome, But not in ulnar neuropathy at the elbow? Muscle Nerve. 2016 Aug;54(2):344. doi: 10.1002/mus.25171. Epub 2016 May 26. No abstract available. PMID 27144462
- [Result] Podnar S, Omejec G. Why do local corticosteroid injections work in carpal tunnel syndrome, but not in ulnar neuropathy at the elbow? Muscle Nerve. 2016 Apr;53(4):662-3. doi: 10.1002/mus.24956. No abstract available. PMID 26506508
- [Result] Bodor M, Rojo-Manaute JM, Podnar S. Reply. Muscle Nerve. 2016 Aug;54(2):344-5. doi: 10.1002/mus.25170. No abstract available. PMID 27144365